CLINICAL TRIAL: NCT00997828
Title: Randomized Comparison of Coronary Artery Bypass Surgery and Everolimus-Eluting Stent Implantation in the Treatment of Patients With Multivessel Coronary Artery Disease (BEST)
Brief Title: Bypass Surgery Versus Everolimus-Eluting Stent Implantation for Multivessel Coronary Artery Disease (BEST)
Acronym: BEST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Problem with recruitment of subjects
Sponsor: Seung-Jung Park (Other)
Collaborators: Abbott Medical Devices (Industry); CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, Chairman,Heart Institute, Asan Medical Center,University of Ulsan,College of Medicine, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008-0272
Record Dates: First submitted 2009-10-18; First posted 2009-10-19 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; stent; coronary artery bypass graft surgery; multivessel coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coronary Artery Bypass

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- everolimus-eluting stent (Experimental): everolimus-eluting stent
  Interventions: Device: everolimus-eluting stent
- coronary artery bypass graft surgery (Active Comparator): coronary artery bypass graft surgery
  Interventions: Procedure: coronary artery bypass graft surgery

INTERVENTIONS:
Device: everolimus-eluting stent — Xience V stent
  Other Names: everolimu-eluting stent
  Arms: everolimus-eluting stent
Procedure: coronary artery bypass graft surgery — coronary artery bypass graft surgery
  Arms: coronary artery bypass graft surgery

SUMMARY:
The purpose of this study is to determine whether the safety and efficacy of coronary stent implantation using Everolimus-Eluting Coronary Stent System (Abbott, Boston Scientific) is not inferior to coronary artery bypass grafting (CABG) for the treatment of patient with multivessel coronary artery disease (CAD).

DETAILED DESCRIPTION:
The primary purpose of the BEST Study is to determine whether the safety and efficacy of coronary stent implantation using everolimus-eluting balloon expandable stents is not inferior to coronary artery bypass grafting for the treatment of multivessel coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of older
* Angiographically confirmed multivessel CAD [critical (>70%) lesions in at least two major epicardial vessels and in at least two separate coronary artery territories (LAD, LCX, RCA)] and amenable to either PCI or CABG.
* Indication for revascularization based upon symptoms of angina and/or objective evidence of myocardial ischemia
* Geographically accessible and willing to come in for required study visits
* Signed informed consent.

Exclusion Criteria:

* Severe congestive heart failure (class III or IV according to NYHA, or pulmonary edema) at the time of enrollment.
* Planned simultaneous surgical procedure unrelated to coronary revascularization (e.g. valve repair/replacement, aneurysmectomy, carotid endarterectomy or carotid stent).
* In-stent restenosis of a target vessel
* Prior CABG surgery
* Prior PCI with stent implantation within 1 year
* Two or more chronic total occlusions in major coronary territories
* Acute ST-elevation MI(Q-wave) within 72 hours prior to enrollment requiring revascularization
* Abnormal creatine kinase (CK > 2x normal) and/or abnormal CK-MB levels and/or elevated Troponin levels at time of randomization
* Previous stroke within 6 months or patients with stroke at more than 6 months with significant residual neurologic involvement, as reflected in a Rankin Score > 1
* Dementia with a Mini Mental Status Examination (MMSE) score of ≤ 20
* Extra-cardiac illness that is expected to limit survival to less than 2 years; e.g. oxygen-dependent chronic obstructive pulmonary disease, active hepatitis or significant hepatic failure, severe renal disease.
* Prior history of significant bleeding (within the previous 6 months) that might be expected to occur during CABG or PCI/DES related anticoagulation.
* Contraindication either CABG or PCI/DES because of a coexisting clinical condition
* Significant leucopenia, neutropenia, thrombocytopenia, anemia, or known bleeding diathesis
* Intolerance or contraindication to aspirin or both clopidogrel and ticlopidine
* Suspected pregnancy. A pregnancy test (urine or serum) will be administered prerandomization to all women not clearly menopausal
* Concurrent enrollment in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 888 (Actual)
Dates: Start 2008-07-28 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
the composite of death, nonfatal myocardial infarction, and ischemia-driven target vessel revascularization (TVR) | at 2 years
  Death includes all cause mortality. MI includes both Q wave and non Q wave, per protocol definition. TVR should be defined by the protocol.

SECONDARY OUTCOMES:
the composite of death, myocardial infarction, and any target vessel revascularization | at 2years
Ischemic MACCE (The composite of death, MI, stroke and ischemia-driven TVR) | at 2 years
MACCE (The composite of death, MI, stroke and any TVR) | at 2 years
the composite of death, MI, and any TVR | at 30 days and yearly to 5 years
ischemic MACE(the composite of death, MI, and any TVR) | at 30 days and yearly to 5 years
MACCE (The composite of death, MI, stroke and ischemia-driven TVR) | at 30 days and yearly to 5 years
ischemic MACCE(The composite of death, MI, stroke and ischemia-driven TVR) | at 30 days and yearly to 5 years
all cause death | at 30 days and yearly to 5 years
cardiac death | at 30 days and yearly to 5 years
myocardial infarction | at 3o days and yearly to 5 years
stroke | at 30 days and yearly to 5 years
ischemic-driven TVR | at 30 days and yearly to 5 years
any target vessel revascularization | at 30 days and yearly to 5 years
any target vessel revascularization or target lesion revascularization | at 30 days and yearly to 5 years
non-target vessel revascularization | at 30 days and yearly to 5 years
stent thrombosis for the percutaneous coronary intervention arm; acute, subacute, and late | at 30 days and yearly to 5 years
analysis segment and in-stent binary restenosis | at 9 months angiographic follow-up
analysis segment and in-stent late loss | at 9 months angiographic follow-up
angina status | at 2 years
Follow-up in-stent, in-segment neointimal hyperplasia volume by IVUS | at 9 months angiographic follow-up
Incidence of stent malapposition, strut fracture, and peri-stent remodeling by IVUS | at 9 months angiographic follow-up
Graft patency in subjects undergoing CABG (defined as: stenosis [DS>50%] in any of the grafts from touch-down to touch-down point) | at 9 months angiographic follow up
Cardiac re-hospitalizations | at 1 years and yearly to 5 years
Quality of life measurements | at 1 year
use of cardiac medications | at 1 year and yearly to 5 years
Dialysis/hemofiltration | at 30 days and yearly to 5 years
Infectious complications | at 30 days
duration of hospitalization related to the target procedure | at every event time
2-year MACE according to the use of FFR-guided multivessel PCI | at 2 years after index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, PhD, Principal Investigator — Department of Medicine, Asan Medical Center, University of Ulsan College of Medicine
Locations (27):
- China (2):
  - Sir Run Run Shaw Hospital, Hangzhou
  - Zhongshan Hospital, Shanghai
- Malaysia (2):
  - National Heart Institue, Kuala Lumpur
  - Sarawak General Hospital, Kuching
- South Korea (22):
  - Gangwon National Univ. Hospital, Chuncheon
  - Keimyung University Dongsan Medical Center, Daegu
  - Yeungnam University Medical Center, Daegu
  - Konyang University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Inje University Ilsan Paik Hospital, Ilsan
  - National Health Insurance Corporation Ilsan Hospital, Ilsan
  - Gachon University Gil Hospital, Incheon
  - Inje University Pusan Paik Hospital, Pusan
  - Pusan National University Yangsan Hospital, Pusan
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Hanyang National University Medical Center, Seoul
  - Inje University Sanggye Paik Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Severance Hospital, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul
  - St.carollo Hospital, Suncheon
  - Ulsan University Hospital, Ulsan
  - Wonju Christian Hospital, Wŏnju
- Siriraj Hospital, Bangkok, Thailand

REFERENCES:
- [Derived] Lee J, Ahn JM, Kim H, Choi Y, Jo S, Kang DY, Kim MJ, Hur SH, Park HJ, Tresukosol D, Kang WC, Kwon HM, Rha SW, Lim DS, Jeong MH, Lee BK, Huang H, Lim YH, Bae JH, Kim BO, Ong TK, Ahn SG, Chung CH, Park DW, Park SJ; BEST Extended Follow-up Study investigators. Long-term outcomes of intravascular ultrasound-guided percutaneous coronary intervention versus coronary artery bypass grafting for multivessel coronary artery disease. Heart. 2025 Sep 11;111(19):918-924. doi: 10.1136/heartjnl-2024-325107. PMID 40368452
- [Derived] Kim H, Kang DY, Ahn JM, Lee J, Choi Y, Hur SH, Park HJ, Tresukosol D, Kang WC, Kwon HM, Rha SW, Lim DS, Jeong MH, Lee BK, Huang H, Lim YH, Bae JH, Kim BO, Ong TK, Ahn SG, Chung CH, Park DW, Park SJ; BEST Extended Follow-Up Study Investigators. Everolimus-Eluting Stents or Bypass Surgery for Multivessel Disease in Diabetics: The BEST Extended Follow-Up Study. JACC Cardiovasc Interv. 2023 Oct 9;16(19):2412-2422. doi: 10.1016/j.jcin.2023.07.028. PMID 37821187
- [Derived] Ahn JM, Kang DY, Yun SC, Ho Hur S, Park HJ, Tresukosol D, Chol Kang W, Moon Kwon H, Rha SW, Lim DS, Jeong MH, Lee BK, Huang H, Hyo Lim Y, Ho Bae J, Ok Kim B, Kiam Ong T, Gyun Ahn S, Chung CH, Park DW, Park SJ; BEST Extended Follow-Up Study Investigators. Everolimus-Eluting Stents or Bypass Surgery for Multivessel Coronary Artery Disease: Extended Follow-Up Outcomes of Multicenter Randomized Controlled BEST Trial. Circulation. 2022 Nov 22;146(21):1581-1590. doi: 10.1161/CIRCULATIONAHA.122.062188. Epub 2022 Sep 19. PMID 36121700
- [Derived] Takahashi K, Serruys PW, Fuster V, Farkouh ME, Spertus JA, Cohen DJ, Park SJ, Park DW, Ahn JM, Onuma Y, Kent DM, Steyerberg EW, van Klaveren D; SYNTAX, BEST, and FREEDOM Trial investigators. External Validation of the FREEDOM Score for Individualized Decision Making Between CABG and PCI. J Am Coll Cardiol. 2022 Apr 19;79(15):1458-1473. doi: 10.1016/j.jacc.2022.01.049. PMID 35422242
- [Derived] Sotomi Y, Onuma Y, Cavalcante R, Ahn JM, Lee CW, van Klaveren D, de Winter RJ, Wykrzykowska JJ, Farooq V, Morice MC, Steyerberg EW, Park SJ, Serruys PW. Geographical Difference of the Interaction of Sex With Treatment Strategy in Patients With Multivessel Disease and Left Main Disease: A Meta-Analysis From SYNTAX (Synergy Between PCI With Taxus and Cardiac Surgery), PRECOMBAT (Bypass Surgery Versus Angioplasty Using Sirolimus-Eluting Stent in Patients With Left Main Coronary Artery Disease), and BEST (Bypass Surgery and Everolimus-Eluting Stent Implantation in the Treatment of Patients With Multivessel Coronary Artery Disease) Randomized Controlled Trials. Circ Cardiovasc Interv. 2017 May;10(5):e005027. doi: 10.1161/CIRCINTERVENTIONS.117.005027. PMID 28495897
- [Derived] Cavalcante R, Sotomi Y, Zeng Y, Lee CW, Ahn JM, Collet C, Tenekecioglu E, Suwannasom P, Onuma Y, Park SJ, Serruys PW. Coronary bypass surgery versus stenting in multivessel disease involving the proximal left anterior descending coronary artery. Heart. 2017 Mar;103(6):428-433. doi: 10.1136/heartjnl-2016-309720. Epub 2016 Sep 20. PMID 27651390
- [Derived] Sotomi Y, Cavalcante R, van Klaveren D, Ahn JM, Lee CW, de Winter RJ, Wykrzykowska JJ, Onuma Y, Steyerberg EW, Park SJ, Serruys PW. Individual Long-Term Mortality Prediction Following Either Coronary Stenting or Bypass Surgery in Patients With Multivessel and/or Unprotected Left Main Disease: An External Validation of the SYNTAX Score II Model in the 1,480 Patients of the BEST and PRECOMBAT Randomized Controlled Trials. JACC Cardiovasc Interv. 2016 Aug 8;9(15):1564-72. doi: 10.1016/j.jcin.2016.04.023. PMID 27491605
- [Derived] Park SJ, Ahn JM, Kim YH, Park DW, Yun SC, Lee JY, Kang SJ, Lee SW, Lee CW, Park SW, Choo SJ, Chung CH, Lee JW, Cohen DJ, Yeung AC, Hur SH, Seung KB, Ahn TH, Kwon HM, Lim DS, Rha SW, Jeong MH, Lee BK, Tresukosol D, Fu GS, Ong TK; BEST Trial Investigators. Trial of everolimus-eluting stents or bypass surgery for coronary disease. N Engl J Med. 2015 Mar 26;372(13):1204-12. doi: 10.1056/NEJMoa1415447. Epub 2015 Mar 16. PMID 25774645